CLINICAL TRIAL: NCT04878198
Title: Comparing the Effectiveness of Physical Exercise and Melatonin Supplement in Treating Sleep Disturbance in Children With ASD: A RCT Study
Brief Title: Treatment of Sleep Disturbance in Children With ASD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Education University of Hong Kong (Other)
Collaborators: Chinese University of Hong Kong (Other); Castle Peak Hospital (Other Government); University of Leicester (Other); United Christian Hospital (Other)
Responsible Party: Principal Investigator, Andy Tse Choi-yeung, Assistant Professor, Education University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RG 21/2019-2020R
Record Dates: First submitted 2021-05-04; First posted 2021-05-07 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Physical Exercise; Sleep Disturbance; Autism Spectrum Disorder; Melatonin Deficiency
Keywords: Autism; Children; Physical exercise; Melatonin; Sleep; Hong Kong; Jogging
MeSH Terms: conditions — Motor Activity; Parasomnias; Autism Spectrum Disorder; Autistic Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Jogging intervention (Experimental): This intervention will be a 10-week jogging program consisting of 50 sessions (5 sessions per week, 30 min per session) in each participating school. The jogging program is confined to morning sessions based on the favourable sleep outcomes from previous study. To counteract the possible influence of natural sunlight exposure, all jogging sessions will be confined to indoor setting. Each session will be conducted in an identical format with 5 minutes of warm-up activities, followed by 20 minutes of jogging (intervention), and 5 minutes of cool-down activities. Participants are instructed to jog at a moderate intensity level. The intensity level of jogging will be measured by heart rate monitor (Polar H1). Meanwhile, questionnaire will be given to the research staff assisting the jogging intervention to assess the adherence of the intervention at T2.
  Interventions: Behavioral: Jogging program
- Melatonin supplement group (Experimental): Participants in this intervention group will undergo a 10-week melatonin supplement intervention period, where melatonin supplement (Natrol®, Chatsworth CA) will be provided 30 minutes before bedtime. The prescription time (i.e. 30 minutes before bedtime) and the dosage of 3mg will be used because these are optimal for most of the participants as suggested by Malow and colleagues. 1 mg and 9 mg are not suggested to ensure the effectiveness of the intervention while preventing the potential daytime sleepiness. Similar to the aforementioned intervention, adherence of the intervention will be assessed at T2.
  Interventions: Drug: Melatonin supplement intervention
- Combination group (Experimental): Participants will receive the jogging program and supplemental melatonin dose with identical format as that in the intervention A and B (e.g., identical duration, identical manpower, identical warm-up and cool-down, identical dose, identical acclimation procedure before the intervention adherence of the intervention for this group will also be assessed at T2.
  Interventions: Behavioral: Jogging program; Drug: Melatonin supplement intervention
- Control group (No Intervention): Participants in the placebo control group will receive no jogging and melatonin supplement dosing activity. However, they will be given a placebo flavored similar to the melatonin supplement (compounded by Pharmacare, Mt. Juliet, NT®). Meanwhile, they will also be required to wear an actigraph to control for their physical activity level at the assessment points (i.e. T1, T2, and T3). They will be expected for following their daily routine without participating in any additional formal physical exercise training program throughout the whole study period (T1-T3). After T3, they will be assisted with jogging program to recognize their contribution as controls.

INTERVENTIONS:
Behavioral: Jogging program — This intervention consists of 50 sessions of morning jogging sessions at moderate intensity level. Each intervention session will be administered by a trained research assistant assisted by student helpers. All the research staff (i.e. student helpers and research assistant) will be required to attend a workshop (see educational plan) to standardize the procedure on implementing the intervention, as well as handling and motivating their ASD partners. Motivation techniques in previous protocol will be used to enhance the compliance rate.
  Arms: Combination group; Jogging intervention
Drug: Melatonin supplement intervention — This intervention is a 10-week melatonin supplement intervention where melatonin supplement will be provided 30 minutes before bedtime.
  Arms: Combination group; Melatonin supplement group

SUMMARY:
This RCT study aims to compare effectiveness physical exercise and melatonin supplement on treating sleep disturbance in children with ASD. A four-arm randomized controlled trial with equal allocation ratio to the three intervention groups (i.e., jogging; melatonin supplement, combine jogging and melatonin supplement) and one placebo-control group will be conducted . Actigraph device and sleep log will be used for sleep assessment. 6-sulfoxymelatonin from 24-h and first morning urinary samples. The investigators will monitor the changes of four sleep parameters (sleep onset latency, sleep efficiency, wake after sleep onset and total sleep duration) and the 24-h and first morning melatonin level throughout the whole study.

DETAILED DESCRIPTION:
Children with ASD are characterized by deficits to some extent - from mild to severe - in social interaction, stereotyped behavior and limited interest. Apart from these core symptoms, sleep disturbance is also commonly found in this population. To cope with sleep problems, medication such as supplemental melatonin is commonly used. Melatonin is the primary hormone produced by the pineal gland for properly timing circadian sleep/wake rhythms to enhance sleepiness during night. Previous research indicated that children with ASD tend to have abnormal melatonin secretion and this may contribute to the abnormal development of sleep-wake cycles. Over the past decade, effect of supplemental melatonin on sleep disturbance treatment has been studied widely in children with autism and the efficacy is well recognized.

Apart from supplemental melatonin, researchers have also explored other intervention strategies that could ameliorate the symptoms of sleep disturbance in children with ASD. One intervention strategy that receives growing attention is physical exercise. Previous studies showed that physical exercise could improve sleep quality in children with ASD. Then it is natural to ask which intervention - physical exercise or melatonin supplement is more effective to promote sleep health in the population. This proposed study aims to compare the effectiveness of three interventions, namely, physical exercise, melatonin supplement and the combination of the two, on treating sleep disturbance among children with ASD via a melatonin mediated mechanism model. Two significant impacts will be expected. First, if the three interventions were equally effective, then physical exercise, which is more naturalistic and brings other health benefits, can be an alternative option for practitioners and parents to treat sleep problems for their patients and children with ASD. Second, if there was a difference between the three interventions on treating sleep problems, it will then inform further research on the relationship between physical exercise, supplemental melatonin and sleep. For example, if the combination was the most effective intervention to ameliorate the sleep disturbance in children with ASD, it would imply the investigators may need to further investigate other factors such as neurological factors (e.g. brain derived neurotrophic factor) or psychological factors (e.g. happiness, motivation) that may play a role on mediating the relationship between physical exercise and sleep. Each participant will attend 3 one-week-long assessments in their respective schools, where the investigators will assess their habitual sleep patterns and endogenous melatonin level before the intervention (T1), in the mid of the study (5 weeks after the commencement of the study) (T2) and after the 10-week intervention (T3). The mid-assessment is valuable to know how much variance in sleep behaviors is accounted by variance in melatonin, as well as to assess the adherence of the interventions.

The findings of this study will allow the investigators to reaffirm if melatonin mediates the relation between physical exercise and changes in sleep quality, which would further strengthen the current limited evidence on the efficacy of physical exercise for sleep problems in children with ASD. The findings of the proposed study will ultimately lead to optimal treatment interventions for sleep disturbance not only in children with ASD, but also in any population suffering from sleep disturbances.

ELIGIBILITY:
Inclusion Criteria:

* age 8 - 12 years
* clinical diagnosis of ASD from a physician or clinical psychologist based on the Diagnostic and Statistical Manual of Mental Disorders, 5th edition, (DSM-5) and confirmed with the Autism Diagnostic Interview- Revised (ADI-R)
* pre-puberty as indicated by Tanner stage I through screening by a physician
* being given an average of 8 hours of sleep per night by their parents over the past 3 months
* parents reported sleep onset delays of 30 minutes of longer on three or more nights per week
* free of psychotropic medications (allergy medications and medications for constipation are allowed)
* non-verbal IQ over 40
* able to perform the requested physical intervention.

Exclusion Criteria:

* with one or co-morbid psychiatric disorders identified with a structured interview based on DSM-5
* with other medical conditions that limit their physical activity participation and sleep (e.g., asthma, seizure, cardiac disease etc)
* with a complex neurologic disorder (e.g., epilepsy, phenylketonuria, fragile X syndrome, tuberous sclerosis)
* participants who are currently meeting physical activity guidelines (more than or equal to 60 minutes of moderate and vigorous physical activity each day).

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 62 (Actual)
Dates: Start 2022-12-02 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Sleep onset latency | 10-week
  Sleep onset latency (length of time taken to fall asleep, expressed in minutes, SOL) will be objectively measured by a GT3X accelerometer
Sleep efficiency | 10-week
  Sleep efficiency (actual sleep time divided by time in bed, expressed as a percent, SE) will be objectively measured by a GT3X accelerometer.
Wake after sleep onset | 10-week
  Wake after sleep onset (length of time they were awake after sleep onset, expressed in minutes, WASO) will be objectively measured by a GT3X accelerometer.
Sleep duration | 10-week
  Sleep duration (total sleep in hours and minutes, SD) will be objectively measured by a GT3X accelerometer.
Parental-assessed sleep quality | 10-week
  Participants' sleep patterns will be logged by their parents using daily sleep diary.
24-h melatonin level | 10-week
  All participants will be instructed to collect a 24-h urine sample. 6-sulfatoxymelatonin, a creatinine-adjusted morning urinary melatonin and representative of melatonin level, will be measured from the sample. The weekend has been chosen to allow the participants to stay at home for sample collection. All urine samples will be collected using 24-h urine bottles containing 0.1L of 0.5M hydrochloric acid as a preservative
First morning void melatonin level | 10-week
  All participants will be instructed to collect the first morning void urine sample. 6-sulfatoxymelatonin, a creatinine-adjusted morning urinary melatonin and representative of melatonin level, will be measured from the sample. All urine samples will be collected using small urine bottles containing 0.1L of 0.5M hydrochloric acid as a preservative

CONTACTS AND LOCATIONS:
Locations (1):
- EdUHK, Hong Kong, China, Hong Kong